CLINICAL TRIAL: NCT01499251
Title: A Phase 1/1b, Open-label Study in Patients With Recurrent Glioblastoma to Assess the Safety and Tolerability of Macitentan in Combination With Dose-dense Temozolomide
Brief Title: Clinical Study on the Safety and Tolerability of Macitentan in Combination With Dose-dense Temozolomide in Patients With Recurrent Glioblastoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Results did not clearly support continuing development in recurrent GBM
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC-055-115
Record Dates: First submitted 2011-12-20; First posted 2011-12-26 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2016-05

CONDITIONS: Glioblastoma
Keywords: glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — macitentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Macitentan (Experimental): Macitentan in combination with dose-dense temozolomide
  Interventions: Drug: Phase 1 Dose Escalation; Drug: Phase 1b; Drug: Ancillary Study

INTERVENTIONS:
Drug: Phase 1 Dose Escalation — Macitentan 30, 60, 90 mg or higher in 30 mg dose increments, given orally, up to 150 mg, then 225 mg, 300 mg and 375 mg, unless otherwise decided by the Safety Monitoring Committee. Dose-dense temozolomide 150 mg/m2 body surface area alternating 1 week on 1 week off.
  Other Names: dose-dense temozolomide; Macitentan
Drug: Phase 1b — Macitentan given orally and daily at doses/schedule determined from the dose escalation period. Dose-dense temozolomide 150mg/m2 body surface area alternating 1 week on 1 week off.
  Other Names: Macitentan; dose-dense temozolomide
Drug: Ancillary Study — Macitentan dosed initially for 8-14 days prior to craniotomy, then treatment interrupted from time of craniotomy until 7 days before start of dose dense temozolomide therapy. dose-dense temozolomide 150 mg/m2 body surface area alternating 1 week on 1 week off.
  Other Names: dose-dense temozolomide; Macitentan

SUMMARY:
This is an open-label, single arm, Phase 1 study to assess the safety and tolerability of macitentan in combination with dose-dense temozolomide in adult patients with recurrent glioblastoma or gliosarcoma. The study is composed of three parts. A Phase 1 Dose Escalation Period with a traditional 3+3 design will determine the maximum tolerated dose of macitentan in combination with dose-dense temozolomide. A Phase 1b Period will expand the safety and tolerability data of two doses of macitentan and dose-dense temozolomide selected from the Dose Escalation Period and explore efficacy. An Ancillary Study will further evaluate the effects of macitentan on biomarkers in brain tumor tissue.

The study is planned to have a minimum duration of 12 months. The study will end when all patients (excluding those prematurely withdrawn or lost to follow-up) in each part of the study have completed a visit at month 12 and 30 days of safety follow-up.

ELIGIBILITY:
Inclusion Criteria

* Histologically confirmed glioblastoma multiforme or gliosarcoma
* Recurrent disease with an:

  * interval of at least 3 months following initial radiotherapy and temozolomide
  * interval of at least 3 weeks between end of surgery for recurrent disease and start of protocol therapy for patients who have undergone surgery for recurrent disease
* KPS 60% or higher
* Adequate bone marrow function Women of childbearing potential must have a negative serum beta-HCG pregnancy test documented within 14 days prior to study initiation.
* Women of childbearing potential must agree to use two reliable methods of contraception from screening and up to 30 days after discontinuation of study treatment.
* Males not naturally or surgically sterile, who have a female partner of childbearing potential, must agree to use two reliable methods of contraception from screening and up to 30 days after discontinuation of study treatment.

Exclusion Criteria

* Histology other than astrocytoma grade IV (GBM or gliosarcoma)
* Tumor foci below the tentorium or or beyond the cranial vault
* Glioblastoma or gliosarcoma disease with leptomeningeal spread
* Patients with a history of any other cancer, unless in complete remission, and off all therapy for that disease for a minimum of 5 years
* Elevated serum aspartate aminotransferase, alanine aminotransferase, or bilirubin (unless there is medical justification for bilirubin elevation, and aspartate aminotransferase, alanine aminotransferase, and alkaline phosphatase are normal)
* Moderate to severe hepatic impairment
* Confirmed systolic blood pressure < 100 mmHg or diastolic blood pressure < 50 mmHg
* History of orthostatic hypotension
* Renal insufficiency or serum creatinine above the normal reference range
* Prior chemotherapy for recurrent glioblastoma with nitrosourea compounds or bevacizumab
* Prior focal radiotherapy
* Severe, active co-morbidity (e.g. cardiac disease; respiratory disease; chronic hepatitis; hematological and bone marrow diseases; severe malabsorption)
* No other active cancer
* No concurrent cytochrome P450 3A4 inducers
* No concurrent strong cytochrome P450 3A4 inhibitors
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2012-01; Primary Completion 2016-01 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose of macitentan in combination with dose-dense temozolomide | Phase I Dose Escalation period (Dose-Limiting Toxicity from Baseline to 28 days for each dose level)

SECONDARY OUTCOMES:
Number of patients with treatment-emergent adverse events (AEs) and serious AEs | Participants will be followed up for the duration of combination treatment, an expected average of 9-12 months.
  for all study periods
Number of patients with AEs leading to premature discontinuation of study treatment | Participants will be followed up for the duration of combination treatment, an expected average of 9-12 months.
  for all study periods
Incidence of treatment-emergent* marked laboratory abnormalities | Participants will be followed up for the duration of combination treatment, an expected average of 9-12 months.
  for all study periods
Number of patients with treatment-emergent ECG abnormalities | Up to 30 days after discontinuation of macitentan
  for all study periods
Change from baseline in vital signs | Up to 30 days after discontinuation of macitentan
  for all study periods: systolic and diastolic blood pressure [supine and standing], average of the two measurements and pulse rate.
Occurrence of at least grade 2 ALT and/or AST elevation | Participants will be followed up for the duration of combination treatment, an expected average of 9-12 months.
  for all study periods

CONTACTS AND LOCATIONS:
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Weathers SP, Rood-Breithaupt J, de Groot J, Thomas G, Manfrini M, Penas-Prado M, Puduvalli VK, Zwingelstein C, Yung WKA. Results of a phase I trial to assess the safety of macitentan in combination with temozolomide for the treatment of recurrent glioblastoma. Neurooncol Adv. 2021 Oct 2;3(1):vdab141. doi: 10.1093/noajnl/vdab141. eCollection 2021 Jan-Dec. PMID 34693288